CLINICAL TRIAL: NCT06056557
Title: Versatility of a Circular Multielectrode Catheter in the Individualized Recognition & Treatment of Atrial Fibrillation and Related Arrhythmias Using Pulsed Field Energy
Acronym: VIRTUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-00978
Record Dates: First submitted 2023-09-06; First posted 2023-09-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation, Paroxysmal or Persistent; Atrial Fibrillation and Flutter; Atrial Flutter Typical
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Non-randomized, interventional clinical study to determine the safety and efficacy in using BWI IRE ablation system in a variety of atrial arrhythmias. All patients will receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional (Experimental): All patients will receive the intervention. That is, all patients will undergo ablation with the experimental catheter (device).
  Interventions: Device: VARIPULSE™ catheter ablation

INTERVENTIONS:
Device: VARIPULSE™ catheter ablation — Subjects will arrive to the electrophysiology laboratory for their ablation procedure and will undergo preparation for the procedure per standard protocol.
  The purpose of an ablation procedure is to scar or destroy the heart tissue causing the atrial fibrillation. The current FDA approved ablation treatments commonly use freezing, radio frequency, or laser, delivered through a catheter that is threaded through blood vessels to the heart, as the energy source to destroy the abnormal tissue.
  The BWI IRE VARIPULSE ablation system used in this study uses a type of energy source called pulse field.
  Pulse field ablation applies ultra-rapid (less than 1 second) electrical fields to the heart muscle to destroy the abnormal tissue. This type of energy is thought to safer and more effective at treating atrial fibrillation.
  ● For a lesion set that cannot be performed using the VARIPULSE catheter technology, a conventional FDA-approved RF ablation

SUMMARY:
The purpose of this pragmatic study is to evaluate the safety, performance and effectiveness of the VARIPULSE catheter technology used in combination with the TRUPULSE™ Generator, and the compatible EAM system (Carto 3D) to treat patients with atrial fibrillation and related arrhythmias during clinically-indicated ablation procedures.

DETAILED DESCRIPTION:
By virtue of its efficiency, safety profile, and potential for improved efficacy in certain patient populations (e.g., thickened atrial tissue of hypertrophic cardiomyopathy (HCM) patients), there is tremendous excitement about the role of pulsed field ablation (PFA) to treat atrial fibrillation and related arrhythmias. However, most PFA clinical trials enroll very selected populations and have highly focused inclusion/exclusion criteria - for example, typically only paroxysmal or persistent atrial fibrillation (AF) patients with upper age criteria are included, other disease states such as HCM are excluded, and typically redo ablation procedures are also excluded. The latter is particularly problematic since redo procedures are quite prevalent in most physicians' clinical practice.

In some sense, the incorporation of these restrictive criteria is not terribly surprising since most of the novel PFA catheters are specifically designed to perform only certain aspects of the AF ablation procedure (e.g., just PVI). That is, when there are more complex substrates (where other types of lesion sets may be needed), it may not be practical to allow a more inclusive criteria for enrollment. Of course, the downside is that the majority of the patients that are eventually treated in clinical practice are not reflected by the enrolled patient population.

The VARIPULSE™ catheter technology is a novel circular catheter with a variable loop design, containing multiple electrodes with individual irrigation pores capable of delivering pulse-field energy.

The Ablation procedure will follow the below sequence:

* Anatomical and voltage mapping of the left and/or right atrium
* To perform this mapping, the VARIPULSE bi-directional catheter or a compatible conventional FDA-approved multi-electrode mapping catheter (e.g., Pentaray, Octaray or Optrell) may be used
* Activation mapping of any-presenting or inducible atrial flutter
* Pulmonary Vein Isolation (PVI) to be achieved in all patients with atrial fibrillation (if not already achieved).
* Confirmation of entrance block with adenosine or isoproterenol challenge
* Additional ablation lesion sets are per the investigator's discretion including:

  * Posterior wall Isolation
  * Regional fractionation clusters
  * Cavo-tricuspid isthmus Line
  * Mitral Isthmus Line
  * Any micro-/macro-reentrant atrial tachycardia's
* As part of the ablation procedure, any safety assessments that are considered important (e.g., EGD, coronary angiography, etc.) may be performed; these data will also be collected.

This study is a prospective, single-center, non-randomized, interventional clinical study to determine the safety and efficacy in using BWI IRE ablation system in a variety of atrial arrhythmias. Subjects will be followed for 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Diagnosed with atrial fibrillation or atrial atypical atrial flutter (typical flutter may also be ablated provided that the typical flutter occurs in addition to atrial fibrillation or atypical flutter; that is, typical flutter as the sole arrhythmia should not undergo PFA).
* Previous surgical or catheter ablation for atrial fibrillation is allowed
* Planned for a catheter ablation procedure
* Able and willing to provide written consent and comply with all testing and follow-up requirements
* Have in place or are planned to receive an implantable loop recorder, pacemaker or defibrillator capable of recording atrial rhythm

Exclusion Criteria:

* Documented "active" left atrial thrombus
* Conditions that preclude the introduction and manipulation of intracardiac catheters: eg, active intracardiac thrombus, myxoma, tumor, a prohibitive interatrial baffle or patch, etc.)
* Previous PCI/MI within the past 1 month
* Active systemic infection or sepsis
* Uncontrolled heart failure - New York Heart Association (NYHA) function class IV.
* History of blood clotting, bleeding abnormalities or contraindication to anticoagulation.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment.
* Women who are pregnant, lactating, or who are of childbearing age and plan on becoming pregnant during this trial.
* Life expectancy or other disease processes likely to limit survival to less than 12 months.
* Currently enrolled in an investigational study evaluating another device, biologic, or drug, that would interfere with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with acute procedural success | up to 12 months post-procedure
  Acute procedural success is defined according to the type of arrhythmia, for example:
  * Entrance block in all targeted PVs for patients treated for atrial fibrillation (Both first and Re-Do)
  * Termination of atrial flutters for patients presenting in atrial flutter.

SECONDARY OUTCOMES:
Percentage of time spent in atrial flutter/fibrillation/tachycardia | up to 12 months post-procedure
  Percentage of time spent in atrial flutter/fibrillation/tachycardia as noted on CIED interrogation.
Percentage of patients with no evidence of atrial fibrillation/flutter or tachycardia of more than 30 seconds of duration | after 3-month blanking period until end of 12 months of follow-up
  The percentage of patients with no evidence of atrial fibrillation/flutter or tachycardia of more than 30 seconds of duration as noted by implantable device after the 3-month blanking period until the end of 12 months of follow-up
Percentage of patients presenting with persistent atrial fibrillation with no evidence of atrial fibrillation/flutter or tachycardia of more than 30 seconds | after 3-month blanking period until end of 12 months of follow-up
  The percentage of patients presenting with persistent atrial fibrillation with no evidence of atrial fibrillation/flutter or tachycardia of more than 30 seconds of duration as noted by implantable device after the 3-month blanking period until the end of 12 months of follow up in patients not taking anti-arrhythmic medications
Percentage of patients who do not report recurrent of symptomatic arrhythmias | after 3-month blanking period until end of 12 months of follow-up
  The percentage of patients who do not report recurrent of symptomatic arrhythmias as noted during telephone or office follow up after the 3-month blanking period until the end of 12 months of follow up
Percentage of patients taking anti-arrhythmic medications with no evidence of atrial fibrillation/flutter or tachycardia of more than 30 seconds | after 3-month blanking period until end of 12 months of follow-up
  The percentage of patients with no evidence of atrial fibrillation/flutter or tachycardia of more than 30 seconds of duration as noted by implantable device after the 3-month blanking period until the end of 12 months of follow up in patients who are taking anti-arrhythmic medications
Percentage of patients not taking anti-arrhythmic medications with no evidence of atrial fibrillation/flutter or tachycardia of more than 30 seconds of duration | after 3-month blanking period until end of 12 months of follow-up
  The percentage of patients with no evidence of atrial fibrillation/flutter or tachycardia of more than 30 seconds of duration as noted by implantable device after the 3-month blanking period until the end of 12 months of follow up in patients who not taking anti-arrhythmic medications
Durability of lesion sets in any patient that undergoes a second procedure | up to 12 months post-procedure
  Durability of lesion sets in any patient that undergoes a second procedure (Block across attempted lines, absence of electrograms in targeted substrate) as measured with 3-d electroanatomic map to assess bidirectional block across ablation lines.
Number of patient emergency room (ER) visits | up to 12 months post-procedure
  Number of patient emergency room (ER) visits
Number of patient Hospitalizations | up to 12 months post-procedure
  Number of patient Hospitalizations
Number of patients requiring cardioversion | up to 12 months post-procedure
  Measured by the actual occurrence of cardioversion procedures
Number of patients who experience repeat ablation | up to 12 months post-procedure
  Number of patients who experience repeat ablation

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data not available/not applicable.